CLINICAL TRIAL: NCT03206203
Title: A Phase II Trial of Atezolizumab (Anti-PDL1) With Carboplatin in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Carboplatin With or Without Atezolizumab in Treating Patients With Stage IV Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Vandana Abramson, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 15136; NCI-2017-01150 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Triple Negative Breast Cancer; Stage IV Breast Cancer; HER2 Negative; Invasive Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — atezolizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (atezolizumab, carboplatin) (Experimental): Patients receive atezolizumab IV over 30-60 minutes and carboplatin IV on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Other: Laboratory Biomarker; Other: Quality-of-Life Assessment
- Arm 2 (atezolizumab, carboplatin) (Experimental): Patients receive carboplatin as in Arm 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may cross-over to Arm 1 upon disease progression.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Other: Laboratory Biomarker; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Atezolizumab — Given by vein
Drug: Carboplatin — Given by vein
Other: Laboratory Biomarker — Correlative study
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well carboplatin with or without atezolizumab works in treating patients with stage IV triple negative breast cancer. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as atezolizumab, may interfere with the ability of tumor cells to grow and spread. Giving carboplatin with atezolizumab may work better in treating patients with stage IV triple negative breast cancer

DETAILED DESCRIPTION:
Primary objective:

To evaluate the efficacy, as measured by progression free survival (PFS) of carboplatin + atezolizumab (using irRECIST) versus carboplatin alone (using RECIST) in patients with triple negative metastatic breast cancer

Secondary objectives:

* To determine overall response rate.
* To evaluate the efficacy, as measured by clinical benefit rate, of carboplatin + atezolizumab (using irRECIST) versus carboplatin (using RECIST) alone in patients with triple negative metastatic breast cancer. Clinical benefit rate is defined as complete response plus partial response plus stable disease for 6 months.
* To determine the duration of response for patients achieving a partial or complete response.
* To evaluate the overall survival (OS) of carboplatin + atezolizumab versus carboplatin alone in patients with triple negative metastatic breast cancer.

TERTIARY OBJECTIVES:

* To perform the following correlative studies from biopsies taken at baseline:

  1. Tumor infiltrating lymphocyte frequency and phenotype (TILs) at baseline
  2. PD-L1 expression from the baseline pre-treatment tissue and at progression lesion, performed by IHC (SP142 clone)
  3. HER2 (IHC, FISH) and ER/PR levels (IHC) from a metastatic site
  4. Perform RNA-seq to determine non-synonymous mutation burden in expressed genes and gene expression to assign a triple negative subtype at baseline for correlations with clinic outcome
  5. Immune phenotyping (IHC) for markers of T cell subsets and activation (CD4, CD8, FoxP3, CD25, Glut1) and exhaustion (PD1, CTLA4) and test feasibility of flow cytometric analyses to include additional markers
* To assess the effect of BRCA mutations on response to the study drugs
* To evaluate the effect of steroids on the efficacy of atezolizumab To assess the prognostic effects of TILs on PFS and CBR in patients receiving atezolizumab

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide informed written consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Clinical stage IV ER, PR, HER2 negative invasive mammary carcinoma, previously documented by histological analysis and that meets the following criteria:
* HER2 negativity is defined as any of the following by local laboratory assessment: In-situ hybridization (ISH) non-amplified (ratio of HER2 to CEP17 < 2.0 or single probe average HER2 gene copy number < 4 signals/cell), or IHC 0 or IHC 1+ (if more than one test result is available and not all results meet the inclusion criterion definition, all results should be discussed with the protocol chair to establish eligibility of the patient)
* ER and PR negativity are defined as =< 5% of cells expressing hormonal receptors via IHC analysis
* Willing to undergo biopsy of a metastatic lesion (in patients with reasonably accessible metastatic lesions such as chest wall, skin, subcutaneous tissue, lymph nodes, bones, peripheral lung, and liver metastases)
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension by RECIST criteria version (v)1.1
* Zero or one prior chemotherapy regimens for metastatic disease
* No prior treatment with carboplatin
* Absolute neutrophil count (ANC) >= 1500/mm^3 (without granulocyte colony-stimulating factor [G-CSF] support within 2 weeks prior to cycle 1, day 1)
* Lymphocyte count >= 500/uL
* Platelet count >= 100,000/mm^3 (without transfusion within 2 weeks prior to cycle 1, day 1)
* Hemoglobin >= 9.0 g/dL

  * Patients may be transfused or receive erythropoietic treatment to meet this criterion
* Calculated creatinine clearance >= 30 mL/min using the Calvert Formula
* Bilirubin =< 2.5 x upper limits of normal if no liver metastases present; serum total bilirubin must be =< 3 x upper limits of normal for patients with Gilbert disease; total bilirubin =< 5 x upper limits of normal if liver metastases present
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) =< 2.5 x upper limits of normal if no liver metastases present; SGOT, SGPT =< 5 x upper limits of normal if liver metastases present
* Alkaline phosphatase =< 2.5 x upper limits of normal if no liver metastases present; alkaline phosphatase =< 5 x upper limits of normal if liver metastases present
* For patients who are not postmenopausal (women) or surgically sterile (absence of ovaries and/or uterus or vasectomy), agreement to remain abstinent or to use two adequate methods of contraception (e.g., condoms, diaphragm, vasectomy/vasectomized partner, tubal ligation), during the treatment period and for at least 30 days after the last dose of study treatment; hormone based oral contraceptives are not allowed on study; postmenopausal is defined as:
* Age >= 60 years
* Age =< 60 years and amenorrheic for 12 months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression; or follicle stimulating hormone and estradiol in the postmenopausal range
* Subjects must complete all baseline screening assessments

Exclusion Criteria:

* CANCER-SPECIFIC EXCLUSION CRITERIA
* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to randomization
* Known central nervous system (CNS) disease, except for treated asymptomatic CNS metastases, provided all of the following criteria are met: measurable disease outside the CNS, only supratentorial metastases allowed (i.e., no metastases to midbrain, pons, medulla, or spinal cord), no evidence of progression or hemorrhage after completion of CNS-directed therapy, no ongoing requirement for dexamethasone as therapy for CNS disease (anticonvulsants at a stable dose are allowed), no stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to randomization
* Leptomeningeal disease
* Uncontrolled tumor-related pain: patients requiring narcotic pain medication must be on a stable regimen at registration; symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to randomization; patients should be recovered from the effects of radiation; there is no required minimum recovery period; asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to randomization
* Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > upper limit of normal [ULN]) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy; patients who are receiving denosumab must discontinue denosumab use and replace it with a bisphosphonate instead while on study; patients receiving a bisphosphonate for skeletal metastases are not excluded and can continue treatment
* Malignancies other than triple negative breast cancer (TNBC) within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, biological therapy) other than the ones specified in the protocol; any other investigational drugs should be discontinued 2 weeks prior to the first dose of study medication
* GENERAL MEDICAL EXCLUSION CRITERIA
* Women only: pregnancy or lactation
* Evidence of significant uncontrolled concomitant disease that in the opinion of the investigator could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
* Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina; patients with a known left ventricular ejection fraction (LVEF) < 40% will be excluded; patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
* Severe infection requiring systemic treatment within 4 weeks prior to randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Major surgical procedure within 4 weeks prior to randomization or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis; placement of central venous access catheter(s) (e.g., port or similar) is not considered a major surgical procedure and is therefore permitted
* History of severe reactions (e.g. allergic, anaphylactic, or other hypersensitivity) to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis; patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study; patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible for this study
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for human immunodeficiency virus (HIV) (testing required prior to registration)
* Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C
* Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible
* Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
* Active tuberculosis
* Receipt of a live, attenuated vaccine within 4 weeks prior to initiation of study drug (cycle 1, day 1 [C1D1]) or anticipation that such a live, attenuated vaccine will be required during the study
* Prior treatment with CD137 agonists, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or IL-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to randomization
* Treatment with systemic corticosteroids or other systemic immunosuppressant medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to cycle 1, day 1, or anticipated requirement for systemic immunosuppressive medications during the trial; patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study; patients with a history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments performed using magnetic resonance imaging (MRI); the use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed
* Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Georgetown University Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Indiana University Health Melvin Bren Simon Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lehmann BD, Abramson VG, Dees EC, Shah PD, Ballinger TJ, Isaacs C, Santa-Maria CA, An H, Gonzalez-Ericsson PI, Sanders ME, Newsom KC, Abramson RG, Sheng Q, Hsu CY, Shyr Y, Wolff AC, Pietenpol JA. Atezolizumab in Combination With Carboplatin and Survival Outcomes in Patients With Metastatic Triple-Negative Breast Cancer: The TBCRC 043 Phase 2 Randomized Clinical Trial. JAMA Oncol. 2024 Feb 1;10(2):193-201. doi: 10.1001/jamaoncol.2023.5424. PMID 38095878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled onto this study at 6 academic medical centers from August 2017 to October 2020.
Groups:
- Arm 2 (Carboplatin): Patients receive carboplatin as in Arm 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may cross-over to Arm 1 upon disease progression.
  Carboplatin: Given by vein
  Laboratory Biomarker: Correlative study
  Quality-of-Life Assessment: Ancillary studies
- Cross-Over: Patients on Arm 2 have the option to cross-over to Arm 1 upon disease progression and receive atezolizumab by IV over 30-60 minutes
Period: Treatment
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin) | Cross-Over
Started | 56 | 50 | 0
Completed | 5 | 2 | 0
Not Completed | 51 | 48 | 0
Not completed — Death | 38 | 26 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — N/A in Follow-Up | 8 | 1 | 0
Not completed — Disease progression | 0 | 1 | 0
Not completed — Refused follow-up | 0 | 1 | 0
Not completed — Cross over to Arm 1 | 0 | 19 | 0
Period: Optional Cross-Over
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin) | Cross-Over
Started | 0 | 0 | 19
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 16
Not completed — Death | 0 | 0 | 14
Not completed — Refused follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin) | Cross-Over | Total
Number analyzed (Participants) | 56 | 31 | 19 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 22 | 16 | 80
  >=65 years | 14 | 9 | 3 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 31 | 19 | 106
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 28 | 18 | 9 | 55
  Unknown or Not Reported | 27 | 13 | 10 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 9 | 3 | 20
  White | 42 | 18 | 13 | 73
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 56 | 31 | 19 | 106

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The PFS is defined as the time from the first day of treatment to the first observation of disease progression (RECIST V1.1) or death of any cause. Those without events were censored at the last follow up. The median PFS time will be estimated using the Kaplan-Meier method with 95% confidence intervals.
Time Frame: Up to 3 years.
Population: Randomized patients received treatments.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 2 (Carboplatin): Patients receive carboplatin as in Arm 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may cross-over to Arm 1 upon disease progression.
  Atezolizumab: Given by vein
  Carboplatin: Given by vein
  Laboratory Biomarker: Correlative study
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin)
Number analyzed (Participants) | 56 | 50
months | 4.1 [2.4 to 7.0] | 2.2 [2.0 to 4.4]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Patient response to treatment was evaluated by RECIST V1.1. The ORR (CR + PR) and corresponding 95% confidence intervals (exact) were estimated among evaluable patients.
Time Frame: Up to 3 years
Population: Randomized patients who received treatments and evaluated for response with evaluanble result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin)
Number analyzed (Participants) | 54 | 45
percentage of participants | 31.5 [21 to 45] | 8.9 [4.0 to 21]

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Patient response to treatment was evaluated by RECIST 1.1. The CBR (CR + PR+stable disease ≥ 6 months) and corresponding 95% confidence intervals (exact) were estimated among evaluable patients.
Time Frame: Up to 3 years
Population: Randomized patients who received treatment and evaluated response with evaluable result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin)
Number analyzed (Participants) | 54 | 45
percentage of participants | 38.9 [27 to 52] | 20.0 [11 to 39]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from CR or PR to progression using RECIST V1.1. The median DOR and corresponding 95% confidence intervals was estimated uisng Kaplan-Meier method.
Time Frame: Up to 3 years
Population: Randomized patients who received treatment and had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin)
Number analyzed (Participants) | 17 | 4
months | 11.6 [7.6 to 17.7] | 14.8 [8.2 to NA] — Too few number of patients to estimate.

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first day of treatment to death. Those alive were censored at the last follow up. The median and OS time and corresponding 95% confidence intervals were estimated using Kaplan-meier method.
Time Frame: Up to 3 years.
Population: Randomized patients who received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin)
Number analyzed (Participants) | 56 | 50
months | 12.6 [10.9 to 19.9] | 7.0 [3.2 to 10.1]

6. Other Pre Specified Outcome: Changes in Gene Expression in Tumor Tissue as Assessed by Ribonucleic Acid-sequencing (RNA-seq)
Description: Statistics will be primarily descriptive.
Time Frame: Baseline and upon disease progression, assessed for up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Assignment of a Triple Negative Subtype in Tumor Tissue as Assessed by Ribonucleic Acid-sequencing (RNA-seq)
Description: Statistics will be primarily descriptive.
Time Frame: Baseline and upon disease progression, assessed for up to 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Define Mutations Present in the Tumors as Assessed by Ribonucleic Acid-sequencing (RNA-seq)
Description: Statistics will be primarily descriptive.
Time Frame: Baseline and upon disease progression, assessed for up to 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Somatic Single Nucleotide Polymorphisms (SNPs) and Structural Variants in Tumor Tissue and Blood as Assessed by Whole Exome Sequencing (WES)
Description: Statistics will be primarily descriptive.
Time Frame: Up to 3 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Status of p53, BRCA1/2, PIK3CA, PTEN, INPP4B and Other Mutations
Description: Statistics will be primarily descriptive.
Time Frame: Up to 3 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Deaths were assessed for up to 3 years. Adverse Events were assessed for an average of 2 years.
Arm/Group | Arm 1 (Atezolizumab, Carboplatin) | Arm 2 (Carboplatin) | Cross-Over
All-Cause Mortality (participants affected / at risk) | 38/56 | 26/50 | 14/19
Serious Adverse Events (participants affected / at risk) | 23/56 | 11/50 | 12/19
Other Adverse Events (participants affected / at risk) | 54/56 | 30/50 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Atezolizumab, Carboplatin) (N=56) | Arm 2 (Carboplatin) (N=50) | Cross-Over (N=19)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 4 (4) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehyration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in left hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombus (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoplysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Disease progression and brain metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Optic Neuritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Altered mental status (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection-E-coli (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Atezolizumab, Carboplatin) (N=56) | Arm 2 (Carboplatin) (N=50) | Cross-Over (N=19)
Limb edema (General disorders) | 4 (4) | 2 (2) | 1 (1)
Flu-Like Symptoms (General disorders) | 3 (3) | 1 (1) | 2 (2)
Chills (General disorders) | 4 (4) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 18 (40) | 14 (31) | 2 (2)
White blood cell decreased (Investigations) | 19 (56) | 14 (27) | 2 (2)
Alanine aminotransferase increased (Investigations) | 14 (16) | 7 (8) | 3 (4)
Creatinine increased (Investigations) | 2 (3) | 3 (3) | 2 (3)
Hemoglobin increased (Investigations) | 3 (9) | 3 (5) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (7) | 5 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (10) | 2 (3) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 15 (32) | 15 (21) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 10 (11) | 9 (11) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (8) | 2 (4) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (7) | 3 (8) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (8) | 6 (6) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (11) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (6) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (10) | 2 (2) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (2) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (10) | 4 (6) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (7) | 5 (5) | 1 (2)
Depression (Psychiatric disorders) | 5 (5) | 2 (2) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 5 (6) | 2 (2)
Hypertension (Vascular disorders) | 3 (7) | 4 (5) | 0 (0)
Hot flashes (Vascular disorders) | 4 (5) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 7 (9) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 3 (4) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 3 (4) | 2 (2) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT03206203/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03206203/ICF_001.pdf